CLINICAL TRIAL: NCT06995053
Title: Image-Guidance With Triggered Beam Hold To Implanted Fiducial Markers or Hypersight for Stereotactic Body Radiotherapy for Prostate Cancer (ILLUSION)
Brief Title: Computed Tomography-Guided Stereotactic Body Radiation Therapy With Intrafraction Motion Monitoring for the Treatment of Localized Prostate Cancer, ILLUSION Trial
Acronym: ILLUSION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0284; NCI-2025-02120 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-06

CONDITIONS: Localized Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (CT-guided SBRT, intrafraction motion monitoring) (Experimental): Patients undergo CT-guided SBRT with intrafraction motion monitoring over 5 fractions every other day, or on consecutive days, if necessary, in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI on study and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: CT-guided Stereotactic Body Radiation Therapy; Other: Intrafraction Motion Monitoring; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Radiation: CT-guided Stereotactic Body Radiation Therapy — Undergo CT-guided SBRT with intrafraction motion monitoring
  Other Names: Computed Tomography-Guided Stereotactic Body Radiation Therapy; CT-guided SBRT
Other: Intrafraction Motion Monitoring — Undergo CT-guided SBRT with intrafraction motion monitoring
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the side effects of computed tomography (CT)-guided stereotactic body radiation therapy (SBRT) with intrafraction motion monitoring and to see how well it works in treating patients with prostate cancer that has not spread to other parts of the body (localized). In CT-guided SBRT, x-ray-based imaging and cone-beam CTs are used to define and localize the area to be treated with SBRT. SBRT is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body (except the brain). The total dose of radiation is divided into smaller doses given over several days. This type of radiation therapy helps spare normal tissue. A recent randomized trial showed that while SBRT is associated with less urinary incontinence and erectile dysfunction than complete surgical removal of the prostate, there are more urinary irritative side effects and more bowel side effects than with surgery. One source of uncertainty in SBRT that may contribute to genitourinary (GU) and gastrointestinal (GI) side effects is the necessity of treating a "margin" of volume around the prostate to account for its movement during SBRT. Intrafraction motion monitoring is any technique or system designed to track the movement of the body and target during fractions of external beam radiation to keep the beam on target. This allows for the patient to be repositioned, if needed, to ensure delivery of the SBRT to only the planned treatment area. CT-guided SBRT with intrafraction motion monitoring may lower GU and GI side effects by allowing tighter margins, as has been demonstrated with magnetic resonance imaging (MRI)-guided SBRT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the acute physician-scored GU toxicity associated with CT-guided SBRT utilizing a 2mm prostate ± seminal vesicles planning target volume (PTV) margin for localized prostate cancer.

SECONDARY OBJECTIVES:

I. To determine the acute physician-scored GI toxicity associated with the intervention.

II. To determine the late physician-scored toxicity associated with the intervention.

III. To determine the patient-reported quality of life outcomes associated with the intervention.

IV. To determine the 5-year biochemical recurrence-free survival (BCRFS) associated with the intervention.

V. To evaluate intrafraction prostate motion using on-board imaging data acquired during this trial in conjunction with prior data, described above.

OUTLINE:

Patients undergo CT-guided SBRT with intrafraction motion monitoring over 5 fractions every other day, or on consecutive days, if necessary, in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI on study and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 1 and 3 months, every 3 months for the first year, every 6 months for a minimum of 5 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, clinically localized adenocarcinoma of the prostate
* No evidence of metastatic disease in lymph nodes above the bifurcation of the renal arteries, or in bones or visceral organs (nodal disease identified on a prostate-specific membrane antigen [PSMA] positron emission tomography [PET]/CT scan below the bifurcation of the renal arteries are amenable)
* Staging workup as recommended by the National Comprehensive Cancer Network (NCCN) on the basis of risk grouping
* Advanced imaging studies (i.e. PSMA PET/CT and fluciclovine PET/CT scan) can supplant a bone scan if performed first
* Age ≥ 18
* Written informed consent obtained from participant or participant's legal representative and ability for participant to comply with the requirements of the study

Exclusion Criteria:

* Patients with neuroendocrine or small cell carcinoma of the prostate
* Patients with any evidence of distant metastases except that evidence of lymphadenopathy below the level of the renal arteries can be deemed locoregional per the discretion of the investigator
* Prior whole gland cryosurgery, high-intensity focused ultrasound (HIFU) or brachytherapy of the prostate
* Prior pelvic radiotherapy
* History of Crohn's Disease, ulcerative colitis, or ataxia telangiectasia
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the participant or the quality of the data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2035-09-01 (Estimated); Study Completion 2036-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute grade ≥ 2 genitourinary (GU) toxicities | From the start of stereotactic body radiation therapy (SBRT) to 90 days post-SBRT
  Will determine physician-scored GU toxicities by the Common Terminology Criteria for Adverse Events, version 5 (CTCAE v5.0) criteria. Rates will be reported descriptively. Point estimates as well as the associated 95% confidence intervals will be reported.

SECONDARY OUTCOMES:
Incidence of acute grade ≥ 2 gastrointestinal (GI) toxicities | From the start of SBRT to 90 days post-SBRT
  Will determine the physician-scored GI toxicities by the CTCAE v5.0 criteria. Rates will be reported descriptively. The analysis of GI toxicity will be stratified for use of hydrogel spacers or not, as these may reduce both acute and late GI toxicity, and by use of nodal radiotherapy or not, if event rate permits this analysis. Additionally, separate analyses of these secondary endpoints stratifying patients by treatment platform and receipt of online adaptive radiotherapy will be performed.
Cumulative incidence of late grade ≥ 2 GU and GI toxicities | Up to 5 years post-SBRT
  Will determine the physician-scored GU and GI toxicities by the CTCAE v5.0 criteria. Will be analyzed using a cumulative incidence framework. The analysis of GI toxicity will be stratified for use of hydrogel spacers or not, as these may reduce both acute and late GI toxicity, and by use of nodal radiotherapy or not, if event rate permits this analysis. Additionally, separate analyses of these secondary endpoints stratifying patients by treatment platform and receipt of online adaptive radiotherapy will be performed.
Change in International Prostate Symptom Score (IPSS) and Expanded Prostate Cancer Index Composite-26 (EPIC-26) score | Baseline to 5 years post-SBRT
  A 15-point or greater increase in IPSS will be considered clinically relevant. Clinically relevant decrement in EPIC-26 domains will be defined as greater than 18, 14, 12, and 24 points for urinary incontinence, urinary irritative or obstructive, bowel, and sexual domains, respectively. Analysis will be performed using a restricted maximum likelihood-based mixed models repeated measures approach. The model will include the fixed categorical effects of treatment, time, and treatment-by-time interaction, as well as the other fixed baseline covariates. An unstructured covariance structure will be used to model the within-patient errors. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom. The analysis of both acute and late changes in the bowel domain of the EPIC instrument will be stratified for use of hydrogel spacers or not, as these may reduce both acute and late GI bowel symptoms.
Biochemical recurrence-free survival | Up to 5 years post-SBRT
  Biochemical recurrence will be defined as serum prostate-specific antigen (PSA) levels that are 2 ng/mL higher than the nadir PSA achieved after SBRT. Will be estimated by the Kaplan-Meier method as well as descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum).
Intrafraction prostate motion | Baseline, at time of SBRT
  Will evaluate intrafraction prostate motion using on-board imaging data acquired during this trial, as well as imaging data from previously treated patients who received computed tomography-guided SBRT. Analysis of imaging data acquired during this study will be descriptive and exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States